CLINICAL TRIAL: NCT06916728
Title: A Post Approval Multicenter 10 Year Follow-up Observational Trial of Marketed Product - MP01 vs. Surgical Standard of Care (SSOC) Used for the Treatment of Joint Surface Lesions of the Knee
Status: Enrolling by invitation | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Collaborators: Cartiheal (2009) Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-0029-1272
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-05

CONDITIONS: Knee Injuries; Joint Surface Knee Lesions
Keywords: Knee cartilage lesions; joint surface lesions of the knee
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Marketed Product - MP01: Subjects who had joint surface lesions of the knee randomized to be treated with Marketed Product - MP01 in the Pivotal study.
  Interventions: Device: Marketed Product - MP01
- Surgical Standard of Care - SSOC: Subjects who had joint surface lesions of the knee randomized to be treated with Surgical Standard of Care (SSOC) - microfracture or debridement in the Pivotal study.
  Interventions: Procedure: Surgical Standard of Care

INTERVENTIONS:
Device: Marketed Product - MP01 — Marketed Product - MP01 was implanted via a mini-arthrotomy or arthrotomy approach, using the designated surgical tools and surgical technique.
  Groups: Marketed Product - MP01
Procedure: Surgical Standard of Care — As no single, current therapy could be used as a single comparator for the treatment of the knee lesions treated in the pivotal study which included focal cartilage lesions on the one hand and moderate knee osteoarthritis on the other, current general practice (e.g., SSOC: Deb and MFx) was used.
  Deb (SSOC) is a common orthopedic surgical procedure that removes damaged cartilage and tissue from the knee. MFx (SSOC) is another common orthopedic surgical procedure that treats knee cartilage defects by creating small holes in the bone beneath the damaged cartilage.
  Groups: Surgical Standard of Care - SSOC

SUMMARY:
The purpose of the study is to support market adoption and global market access via collection of long-term effectiveness, safety, and radiographic data. The primary hypothesis is that Marketed Product (MP01) retains its superiority over Surgical Standard of Care (SSOC) at 7 years in term of mean improvement in the overall Knee Injury and Osteoarthritis Outcome Score (KOOS).

DETAILED DESCRIPTION:
This is a post approval, multicenter, prospective, comparative, non blinded 10-year follow-up observational study of Marketed Product - MP01 vs SSOC used for the treatment of joint surface lesions of the knee. Up to 12 sites in the United States (US) and outside of the US (OUS) that participated in the pivotal study "A Prospective Multicenter Open-label Randomized Controlled Trial of Marketed Product - MP01 vs. Surgical Standard of Care (SSOC) for the Treatment of Joint Surface Lesions of the Knee" (Marketed Product - MP01 vs. SSOC) will enroll up to 170 subjects who participated in the pivotal study and were not withdrawn due to the index knee requiring a unicompartmental or total knee arthroplasty. Enrolled subjects will be followed up to an additional 5 years post pivotal study procedure. As randomization was 2:1 in the pivotal study, the expected number of Marketed Product - MP01 and SSOC subjects enrolled into this study are approximately 114 and 56, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Participated in the pivotal study.
2. Must be physically and mentally willing and able to comply with the follow-up schedule.
3. Signed and dated the IEC/IRB approved Informed Consent Form and HIPPA (if applicable).

Exclusion Criteria:

1. Withdrawn from the pivotal study due to index knee requiring a unicompartmental or total knee arthroplasty.
2. Chemotherapy in the past 12 months.
3. Participation in other clinical trials involving knee procedures.
4. Vulnerable individual including prisoners (i.e., unable to fully understand all aspects of the study that are relevant to the decision to participate or could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 170 subjects who had joint surface lesions of the knee, participated in the pivotal study and consent to continue follow-up will be enrolled.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2030-02-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) at 7 Years | Baseline and 7 years
  Long-term effectiveness of Marketed Product - MP01 compared to SSOC measured by change in baseline to year 7 in overall KOOS (mean of Pain, Symptoms, Quality of Life (QOL), Function in Daily Living (ADL) and Sports subscales) in subjects treated with Marketed Product - MP01 vs SSOC. Baseline is defined as the pivotal study screening visit.
  Overall scores are converted to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no knee problems (i.e., a lower score is a worse outcome, and high score is a better outcome).

SECONDARY OUTCOMES:
Safety of Marketed Product - MP01 vs SSOC: Time to Event of Secondary Invasive Interventions (excluding intra-articular injections) | up to 10 years
  Kaplan-Meier survival estimates will be used to estimate time to secondary invasive intervention (open procedure, mini open procedure, arthroscopic procedure, including implant removal and conversion to knee arthroplasty) excluding intra-articular injections.
Safety of Marketed Product - MP01 vs SSOC: Time to Event of Secondary Invasive Interventions (including intra-articular injections) | up to 10 years
  Kaplan-Meier survival estimates will be used to estimate time to secondary invasive intervention (open procedure, mini-open procedure, arthroscopic procedure, including implant removal and conversion to knee arthroplasty) including intra-articular injections.
Safety of Marketed Product - MP01 vs SSOC: Cumulative Incidence Rate | up to 10 years
  Cumulative incidence rate up to 10 years of secondary invasive interventions (open procedure, mini-open procedure, arthroscopic procedure, including implant removal and conversion to knee arthroplasty) including intra-articular injections.
Change from Baseline in Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) at 7 Years | Baseline and 7 years
  KOOS evaluates both short and long-term consequences of knee injury and contains 42 items including 5 subscales (pain, other symptoms, QOL, ADL, and sports).
  Subscale scores are converted to a 0-100 scale to determine the Overall score, with 0 representing extreme knee problems and 100 representing no knee problems (i.e., a lower score is a worse outcome, and high score is a better outcome).
Change from Baseline in Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) at 10 Years | Baseline and 10 years
  KOOS evaluates both short and long-term consequences of knee injury and contains 42 items including 5 subscales (pain, other symptoms, QOL, ADL, and sports).
  Subscale scores are converted to a 0-100 scale to determine the Overall score, with 0 representing extreme knee problems and 100 representing no knee problems (i.e., a lower score is a worse outcome, and high score is a better outcome).
Change from Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Subscales at 7 Years | Baseline and 7 years
  KOOS evaluates both short and long-term consequences of knee injury and contains 42 items including 5 subscales (pain, other symptoms, QOL, ADL, and sports). Each item has five possible answer options scored from 0 (no problems) to 4 (extreme problems), and each of the five subscales is calculated as the sum of the associated items. Scores are converted to a 0-100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., best outcome).
Change from Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Subscales at 10 Years | Baseline and 10 years
  KOOS evaluates both short and long-term consequences of knee injury and contains 42 items including 5 subscales (pain, other symptoms, QOL, ADL, and sports). Each item has five possible answer options scored from 0 (no problems) to 4 (extreme problems), and each of the five subscales is calculated as the sum of the associated items. Scores are converted to a 0-100 scale, with 0 representing extreme knee problems (i.e., worse outcome) and 100 representing no knee problems (i.e., best outcome).
Change from Baseline in Tegner Activity Scale Score at 7 Years | Baseline and 7 years
  The Tegner Activity Scale assesses the level of work and sports-based activity prior to injury and level of activity post injury that can be documented on a numerical scale. It is a one- item questionnaire that is scored on an 11-item scale (0 to 10) based on the patient's reported level of activity/work. A level of 0 indicates the worst outcome while a level of 10 represents the best outcome.
Change from Baseline in Tegner Activity Scale Score at 10 Years | Baseline and 10 years
  The Tegner Activity Scale assesses the level of work and sports-based activity prior to injury and level of activity post injury that can be documented on a numerical scale. It is a one- item questionnaire that is scored on an 11-item scale (0 to 10) based on the patient's reported level of activity/work. A level of 0 indicates the worst outcome while a level of 10 represents the best outcome.
Change from Baseline in Total 2000 International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score at 7 Years | Baseline and 7 years
  The IKDC Subjective Knee Evaluation Form assesses the subject's opinion of their knee across 3 domains: symptoms (7 items), sports activity (2 items), and knee function (2 items; note: 'function prior to knee injury' is not included in the overall score). Responses vary for each item. The sum of all items is converted to a scale of 0 to 100, where 100 represents no limitation with activities & absence of symptoms (i.e., the best outcome) and 0 represents the worst outcome.
Change from Baseline in Total 2000 International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score at 10 Years | Baseline and 10 years
  The IKDC Subjective Knee Evaluation Form assesses the subject's opinion of their knee across 3 domains: symptoms (7 items), sports activity (2 items), and knee function (2 items; note: 'function prior to knee injury' is not included in the overall score). Responses vary for each item. The sum of all items is converted to a scale of 0 to 100, where 100 represents no limitation with activities & absence of symptoms (i.e., the best outcome) and 0 represents the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Andrews, Study Chair — Smith & Nephew, Inc.; Galit Reske, Study Chair — Smith & Nephew, Inc.
Locations (8):
- Horizon Clinical Research, La Mesa, California, United States
- AZ Monica, Antwerp, Belgium
- Hadassah Medical Center, Jerusalem, Israel
- Italy (2):
  - Humanitas Gavazzeni, Bergamo
  - Istituto Clinico Humanitas, Milan
- County Hospital Timis Othopedy and Trauma Clinic II, Timișoara, Romania
- Serbia (2):
  - Institut za Ortopedsko hiruske Bolesti "Banjica", Belgrade
  - Klinika Orto MD, Novi Sad

IPD SHARING:
Plan to Share IPD: No